CLINICAL TRIAL: NCT07307248
Title: A Randomized Controlled Trial To Evaluate Early (2-Week) vs. Standard (4-Week) Metal Stent Removal Following Endoscopic Ultrasound Guided WON Drainage.
Brief Title: To Evaluate Early (2-Week) vs. Standard (4-Week) Metal Stent Removal Following Endoscopic Ultrasound Guided WON Drainage
Acronym: STEP1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Mohan Ramchandani, DIRECTOR , INTERVENTIONAL ENDOSCOPY, Asian Institute of Gastroenterology, India
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STEP1
Record Dates: First submitted 2025-12-13; First posted 2025-12-29 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Walled Off Necrosis
Keywords: Early LAMS removal

STUDY DESIGN:
Intervention Model Description: Two-arm parallel randomized controlled trial comparing early (2-week) versus standard (4-week) LAMS removal strategies in patients with walled-off pancreatic necrosis (WON).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Stent Replacement Arm (2-Week LAMS Removal + DPT Placement) (Experimental): Participants in this arm will undergo early removal of the lumen-apposing metal stent (LAMS) at 2 weeks after initial endoscopic drainage for walled-off pancreatic necrosis (WON). Following LAMS removal, a double-pigtail plastic stent (DPT) will be placed across the transmural tract to maintain drainage and reduce the risk of recurrent pancreatic fluid collection (PFC). Patients will undergo follow-up imaging at 3, 6, and 12 months to assess recurrence, complications, and need for reintervention.
  Interventions: Procedure: Standard LAMS Removal with Double-Pigtail Plastic Stent
- Standard Stent Replacement Arm (4-Week LAMS Removal without DPT) (Active Comparator): Participants in this arm will undergo standard removal of the LAMS at 4 weeks after initial endoscopic drainage for walled-off pancreatic necrosis (WON). Patients will be followed at 3, 6, and 12 months to assess recurrence of pancreatic fluid collection (PFC), complications, and reintervention rates.
  Interventions: Procedure: Standard LAMS Removal without DPT

INTERVENTIONS:
Procedure: Standard LAMS Removal with Double-Pigtail Plastic Stent — In the early stent removal arm, LAMS will be removed at 2 weeks followed by placement of a double-pigtail plastic stent (DPT).
  Other Names: EARLY
  Arms: Early Stent Replacement Arm (2-Week LAMS Removal + DPT Placement)
Procedure: Standard LAMS Removal without DPT — In the standard arm, LAMS will be removed at 4 weeks.
  Arms: Standard Stent Replacement Arm (4-Week LAMS Removal without DPT)

SUMMARY:
In adults with walled-off pancreatic necrosis (WON) undergoing endoscopic ultrasound (EUS)-guided transluminal necrosectomy, does early removal of the lumen-apposing metal stent (LAMS) (at 2 weeks or immediately after the last necrosectomy) with placement of a double-pigtail plastic stent (DPT), compared to delayed LAMS removal at 4 weeks without a DPT, result in a lower rate of pancreatic fluid collection (PFC) recurrence or need for reintervention over 12 months.

DETAILED DESCRIPTION:
Management of walled-off pancreatic necrosis (WON) following acute pancreatitis has been transformed by the use of endoscopic ultrasound (EUS)-guided transluminal drainage with a lumen-apposing metal stent (LAMS). The LAMS provides a large-caliber conduit for drainage and allows for direct endoscopic necrosectomy, leading to faster resolution of collections and reduced need for surgical intervention. However, the optimal timing for LAMS removal remains uncertain.

Prolonged retention of LAMS has been associated with several adverse events, including delayed bleeding due to vascular erosion, buried-stent syndrome, stent migration, and tissue hyperplasia at the tract site. Conversely, premature removal of the stent may lead to incomplete drainage, persistent or recurrent pancreatic fluid collections (PFCs), and the need for repeat interventions. Therefore, determining the ideal balance between minimizing stent-related complications and preventing recurrence is a key clinical challenge.

Early removal of the LAMS-either 2 weeks after insertion or immediately after the last necrosectomy session-may reduce the risk of delayed bleeding and other metal stent-related complications. However, to maintain tract patency and allow residual drainage, placement of a prophylactic double-pigtail plastic stent (DPT) at the time of LAMS removal has been proposed. The DPT provides a smaller but stable drainage channel that may prevent premature tract closure and recurrence of fluid collections.

This randomized controlled trial aims to rigorously test whether early LAMS removal combined with DPT placement offers better long-term outcomes compared to standard 4-week LAMS removal without DPT. The results are expected to provide evidence-based guidance on optimizing stent management in patients with WON undergoing endoscopic necrosectomy, balancing efficacy with safety.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Patients with walled-off pancreatic necrosis (WON) undergoing endoscopic ultrasound-guided drainage with lumen-apposing metal stent (LAMS)
* Radiological resolution of the pancreatic fluid collection ≥70% at 2 weeks after index endoscopic drainage, assessed on cross-sectional imaging (CT or MRI)

Exclusion Criteria:

* Presence of chronic pancreatitis
* Pancreatic malignancy (suspected or confirmed)
* Incomplete endoscopic necrosectomy or persistent large necrotic debris on imaging at 2 weeks after drainage
* Occurrence of major procedure-related adverse events within the first 2 weeks, including:
* Clinically significant bleeding
* Infection requiring additional intervention
* Stent migration
* Inability or unwillingness to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Estimated)
Dates: Start 2025-12-25 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence of Pancreatic Fluid Collection (PFC) | 12 months after initial drainage procedure
  Recurrence is defined as the redevelopment of a symptomatic pancreatic fluid collection confirmed on imaging (CT or MRI) after initial resolution following endoscopic drainage and lumen-apposing metal stent (LAMS) removal. The recurrence rate will be compared between the early LAMS removal + double-pigtail plastic stent (DPT) group and the standard 4-week LAMS removal group.

SECONDARY OUTCOMES:
Recurrence of Pancreatic Fluid Collection at 3 and 6 Months | 3 months and 6 months after the initial drainage procedure
  Incidence of PFC recurrence confirmed by imaging (CT/MRI) or symptomatic relapse within 3 and 6 months of the index drainage procedure. Comparison will be made between the early LAMS removal + DPT group and the standard 4-week LAMS removal group.
Stent-Related Adverse Events | Up to 12 months post-procedure
  Incidence of complications directly related to LAMS or DPT placement, including migration, occlusion, infection, or buried stent syndrome.
Need for Reinterventions | Within 12 months after stent removal
  Proportion of patients requiring additional interventions for pancreatic collection management, such as repeat endoscopic drainage, necrosectomy, percutaneous drainage or surgical necrosectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Deepak L Jha, (Medical Gastroenterology), Principal Investigator — Asian Institute of Gastroenterology, Hyderabad
Locations (1):
- Asian Institute of Gastroenterology, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because data sharing is not planned for this study.

REFERENCES:
- [Result] Zeng Y, Yang J, Zhang JW. Endoscopic transluminal drainage and necrosectomy for infected necrotizing pancreatitis: Progress and challenges. World J Clin Cases. 2023 Mar 26;11(9):1888-1902. doi: 10.12998/wjcc.v11.i9.1888. PMID 36998953